CLINICAL TRIAL: NCT00370630
Title: Intravitreal Avastin Versus Intravitreal Avastin and Triamcinolone in Central Retinal Vein Occlusion(CRVO)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8544
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Retinovascular Disease
Keywords: CRVO; Intravitreal Avastin; Intravitreal triamcinolone
MeSH Terms: interventions — Bevacizumab; Triamcinolone

INTERVENTIONS:
Drug: Avastin (Bevacizumab) and triamcinolone

SUMMARY:
In this study we intend to evaluate and compare the outcomes of intravitreal avastin versus avastin and triamcinolone on improving the visual acuity and macular edema and late complications of CRVO like NVI and NVG.

DETAILED DESCRIPTION:
Central retinal vein occlusion (CRVO) is a common retinal vascular disorder with potentially complications like reduced vision resulting from extensive intraretinal hemorrhage, retinal ischemia and persistent macular edema and neovascular glaucoma secondary to iris neovascularization. Macular edema is a common cause of severe visual loss in both branch retinal vein occlusion (BRVO) and central retinal vein occlusion (CRVO). Natural history data indicate that CRVO patients presenting with poor visual acuity (_20/200) have an 80% chance of being left with visual acuity less than 20/200 at final visit, whether the CRVO is ischemic or nonischemic at presentation. Treatments that target the secondary effects of venous occlusion, such as grid laser photocoagulation for macular edema and prophylactic panretinal laser photocoagulation for nonperfused CRVO, were shown to be ineffective in improving visual acuity in the Central Vein Occlusion Study (CVOS). Although panretinal photocoagulation is advocated for reducing the risk of neovascular glaucoma in patients with ischemic CRVO, recent clinical trials have failed to demonstrate any significant benefit with laser photocoagulation in the treatment of macular edema due to CRVO. A number of other treatment options are sometimes used in cases of CRVO, such as oral corticosteroids, intravitreal steroids, vitrectomy, hemodilution, intravitreal tissue plasminogen activator, hyperbaric oxygen, and laser or surgical chorioretinal anastomosis. Studies demonstrating the effectiveness of these treatments are inconclusive, although some benefits have been suggested in recent reports. In recent studies the benefit of antiVEGF agents in improving the macular edema due to CRVO have been shown. In this study we are going to compare the effect of intravitreal antiVEGF (Avastin) with combination of Avastin and Triamcinolon in improving the visual acuity and macular thickness in patients with recent (Less than 6 months) CRVO.

ELIGIBILITY:
Inclusion Criteria:

* CRVO with duration less than 6 months

Exclusion Criteria:

* vision less than 20/320 and vison more than 20/50
* history of galucoma and diabetic retinopathy
* previous laser or intravitreal treatment
* any media opacity that prevents funduscopy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-08; Study Completion 2007-02

PRIMARY OUTCOMES:
Best corrected visual acuity
Macular thickness by OCT

SECONDARY OUTCOMES:
Incidence of NVI

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Moradian, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Siamak Moradian, MD, Tehran, Tehran Province, Iran